CLINICAL TRIAL: NCT03497728
Title: Detection of Microdeletions in the Azoospermia Factor (AZF) Regions on the Human Y Chromosome in Infertile Male Patients
Brief Title: Detection of Microdeletions in the Azoospermia Factor (AZF) Regions in Infertile Male Patients
Status: Terminated | Type: Observational
Why Stopped: halted prematurely
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Collaborators: Anhui Provincial Hospital (Other Government); Tang-Du Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: KYXM-201802
Record Dates: First submitted 2018-03-13; First posted 2018-04-13 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-02

CONDITIONS: Azoospermia or Severe Oligozoospermia
MeSH Terms: conditions — Azoospermia; Oligospermia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood is collected in the morning from each patient and then stored at -20℃. Blood specimen is sent to the Lab in Jabrehoo for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study, we used Multiplex ligation-dependent probe amplification and next-generation sequencing technology to detect AZF microdeletion types accurately in selected genetic locus, and made correlation analysis with clinical treatment results.

DETAILED DESCRIPTION:
Infertility has plagued more than 10% of the world's couples of childbearing age, of which male factors account for half. There are many causes of male infertility, including infection, genital malformations, immune dysfunction, varicocele, erectile dysfunction, drug side effect and chromosomal abnormality. Microdeletion of Azoospermia factor (AZF) in the long arm of the Y chromosome is one of the main genetic factors leading to dyszoospermia. The incidence of AZF microdeletions is 2%~19.4% among male infertile patients in Asia, which is related to the inclusion criteria, STS site selection, population and genetic background.

At present, there are large numbers of studies on AZF microdeletions in male infertility, and provide rich information on male infertility. However, as the main means of detection is multiplex PCR-capillary electrophoresis method, which usually detects sequence-tagged sites(STS) such as AZFa-sY84，sY86，AZFb-sY127，sY134，AZFc- sY1191, sY1291, sY1189,sY254 and sY255, information on other loci is still lacking.

In addition, the shortcomings of this method include false positive and false negative results caused by fuzzy electrophoresis strip or pollution and the presence of high repetition and a large number of palindrome in complex AZF region. Because some microdeletions can't be detected it is difficult to make an accurate judgement on the fertility of the patients.

This study will use Multiplex ligation-dependent probe amplification and NGS method to improve the detection rate of AZF microdeletion, and analyze the microdeletion data and the patient's fertility results, so as to improve genetic counseling. A total of 5000 male infertility patients will be enrolled. At least 1000 parents and 1000 normal fertile men will be asked to donate their peripheral blood for DNA.

In addition, in patients with azoospermia or severe oligozoospermia, the overall deletion rate of AZF is about 8.77% (1.75%-24.70%), so there are other unknown genetic factors leading to azoospermia or severe oligozoospermia. This study will also try to make a preliminary study of these factors.

ELIGIBILITY:
Inclusion Criteria:

-Male patients diagnosed with azoospermia and severe oligozoospermia.

Exclusion Criteria:

1. Klinefelter Syndrome ;
2. Structural chromosome aberrations；
3. Obstructive anspermia;
4. Male infertility caused by endocrine factors;
5. Do not meet requirements for acquisition, processing and preservation of samples；
6. After sampling, it doesn't conform to the standard of quality control, or other experimental conditions that don't meet the test requirement；
7. Unable to obtain patient history;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male patients diagnosed with azoospermia and severe oligozoospermia.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
frequency of mirodeletion | through study completion, an average of 1 year
  The propotion of azoospermia patients with AZF mirodeletion

CONTACTS AND LOCATIONS:
Overall Officials: Yueqiu Tan, Study Chair — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China